CLINICAL TRIAL: NCT01087866
Title: Metformin Versus Insulin in the Treatment of Gestational Diabetes Mellitus: a Randomized Controlled Study
Brief Title: Metformin Versus Insulin in the Treatment of Gestational Diabetes Mellitus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Ijas Hilkka, MD, Dept. Obstetrics and Gynecology, Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 070471
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Gestational diabetes mellitus; treatment; metformin
MeSH Terms: conditions — Diabetes, Gestational | interventions — Metformin; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Experimental)
  Interventions: Drug: Metformin
- Insulin (Active Comparator)
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Metformin
  Arms: Metformin
Drug: Insulin
  Arms: Insulin

SUMMARY:
The purpose of this study is to determine if metformin therapy prevents fetal macrosomy in gestational diabetes mellitus to the same extent as insulin therapy.

ELIGIBILITY:
Inclusion Criteria:

* gestational diabetes mellitus diagnosed between 12-34 pregnancy weeks if normoglycemia is not reached with diet

Exclusion Criteria:

* hypertension with pharmacological treatment or preeclampsia
* multiple pregnancy
* liver or kidney disease

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2005-06; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Percentage of fetal macrosomy

CONTACTS AND LOCATIONS:
Overall Officials: Hilkka Ijas, MD, Principal Investigator — Oulu University Hospital; Tytti Raudaskoski, MD,PhD, Study Director — Oulu University Hospital; Marja Vaarasmaki, MD, PhD, Study Chair — Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Finland

REFERENCES:
- [Derived] Ijas H, Vaarasmaki M, Morin-Papunen L, Keravuo R, Ebeling T, Saarela T, Raudaskoski T. Metformin should be considered in the treatment of gestational diabetes: a prospective randomised study. BJOG. 2011 Jun;118(7):880-5. doi: 10.1111/j.1471-0528.2010.02763.x. Epub 2010 Nov 18. PMID 21083860